CLINICAL TRIAL: NCT00082225
Title: Administration of LMP2a-Specific Cytotoxic T-Lymphocytes Following CD45 Antibody to Patients With Relapsed EBV-Positive Hodgkin's or Non-Hodgkin's Lymphoma
Brief Title: LMP2a-Specific Cytotoxic T-Lymphocytes, Lymphoma (ACDAL)
Acronym: ACDAL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14424-ACDAL; ACDAL (Other: Baylor College of Medicine)
Record Dates: First submitted 2004-05-03; First posted 2004-05-05 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: Hodgkins; Non-Hodgkins; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBV specific T cells (Experimental): Patients receiving CTLs as therapy for relapsed Lymphoma or who are at high risk for relapse or patients receiving CTLs as adjunctive therapy following autologous or syngeneic transplant.
  A fixed dose of CD45 MAb (400ug/kg over 4 hours daily times 4 given over 2 daily IV infusions) will be used.
  Interventions: Biological: CD45 antibodies; Biological: EBV specific T cells

INTERVENTIONS:
Biological: CD45 antibodies — The antibody solution is administered by a syringe pump in incremental doses, 0.2-0.8 mg in the first hour and up to 10 mg/hr thereafter, for a maximum infusion time of 8 hrs.
Biological: EBV specific T cells — The following dose levels will be evaluated: Each patient will receive 1 injection, according to the following dosing schedules:
  2 x 10e7 cells/m2 5 x 10e7 cells/m2
  1 x 10e8 cells/m2

SUMMARY:
Patients have a type of cancer called Hodgkin's lymphoma or non-Hodgkin's lymphoma, which has come back or not gone away or is at high risk for coming back after treatment, including the best treatment investigators know for this disease. Investigators are asking the patient to volunteer to be in a research study using a new experimental therapy consisting of special immune system cells called LMP2 specific cytotoxic T lymphocytes in combination with a special protein called a monoclonal antibody.

Some patients with Hodgkin or non-Hodgkin Lymphoma show evidence of infection with the virus that causes infectious mononucleosis Epstein Barr virus (EBV) before or at the time of their diagnosis of the lymphoma. EBV is found in the cancer cells of up to half the patients with lymphoma, suggesting that it may play a role in causing lymphoma. The cancer cells infected by EBV are able to hide from the body's immune system and escape destruction. Investigators want to see if special white blood cells, called T cells, that have been trained to kill EBV infected cells can survive in the blood and affect the tumor.

The investigators have used this sort of therapy to treat a different type of cancer that occurs after bone marrow and solid organ transplant called post transplant lymphoma. In this type of cancer the tumor cells have 9 proteins made by EBV on their surface. They grew T cells in the laboratory that recognized all 9 proteins and were able to prevent and treat post transplant lymphoma. However in Hodgkin disease and non-Hodgkin Lymphoma the tumor cells only express 2 EBV proteins. In a previous study investigators made T cells that recognized all 9 proteins and gave them to patients with Hodgkin disease. Some patients had a partial response to this therapy but no patients had a complete response. Investigators think one reason may be that many of the T cells reacted with proteins that were not on the tumor cells. They are now trying to find out if they can improve this treatment by growing T cells that only recognize one of the proteins expressed on Lymphoma cells called LMP-2. These special T cells are called LMP-2 specific cytotoxic T-lymphocytes (CTLs).

In this study investigators also are trying to see if they can improve these results by treating patients first with a special protein called an antibody and then giving the EBV specific T cells. The reason for doing this is that EBV specific T cells have worked very well in bone marrow transplant patients to prevent and treat EBV cancers. These patients have very few of their own immune cells when they are given the trained T cells and therefore there is a lot of space for the trained cells to grow. Investigators hope that they can improve the effect of the trained T cells in Hodgkin disease and non-Hodgkin Lymphoma patients by first temporarily removing the patient's own T cells before giving the trained cells.

DETAILED DESCRIPTION:
Investigators first tested a biopsy of the tumor that has already been done to see if the tumor cells are EBV positive. They then got permission to take up to 60ml (12 teaspoonfuls) of blood from the patient or their donor on one or two occasions and used this blood to grow T cells in the laboratory. They first grew a special type of cell called dendritic cells stimulate the T cells and put a specially produced human virus (adenovirus) that carries the LMP-2a gene into the dendritic cells. These dendritic cells were then treated with radiation so they could not grow. They were then used to stimulate T cells. This stimulation trained the T cells to kill cells with LMP-2a on their surface. Investigators then grew these LMP-2a specific CTLs by more stimulation with EBV infected cells (which were made from the patient's blood or their donor's blood by infecting them with EBV in the laboratory). The investigators also put the adenovirus that carries the LMP2 gene into these EBV infected cells to increase the amount of LMP2 that these cells have. Again, these EBV infected cells were treated with radiation so they could not grow. Once sufficient numbers of T cells were made, investigators tested them to make sure they kill cells with LMP2a on their surface. These cells are now ready to give to the patient if they agree to being on this study.

Investigators also took up to 500 ml (2 1/2 cups) of extra blood from the patient or their donor, which were frozen. In case the patient's own cells do not recover as expected after the antibody and cell infusions, these cells can be thawed and given back to the patient.

If the patient agrees to this treatment they will get treated with the CD45 antibodies for 4 days in a row and then 2-3 days later get a dose of LMP2 specific CTLs.

The CD45 antibodies will be given to the patient through a vein for 6-8 hours and monitored for at least 6 hours after the infusion. After the infusion The patient will be checked for the levels of CD45 in the blood at 24 hours (optional) and/or at 48-72 hours after the last infusion to check the level is low enough to give the patient the CTLs.

The CTLs will be thawed and injected through a central line, if the patient has one, or through a vein in their arm over 10 minutes, after pretreatment with Tylenol and Benadryl. We will then monitor them in clinic for 4 hours after the injection.

All of the treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or the Methodist Hospital. We will follow the patient in the clinic after the CTL injection. If there is a reduction in the size of the lymphoma on CT or MRI scans as assessed by a radiologist, they can receive up to six additional doses of the T cells if they wish.

ELIGIBILITY:
Inclusion Criteria:

* Any patient, regardless of age or sex, with EBV-positive Hodgkin's or non-Hodgkin lymphoma, regardless of the histological subtype or EBV-associated T/NK cell Lymphoproliferative disease. This includes patients in second or subsequent relapse including post autologous or syngeneic stem cell transplant (or with active disease or in first relapse if immunosuppressive chemotherapy contraindicated or if the patient has relapsed multiple times and is currently in remission but has a high risk of relapse). (group A) OR Patients who have relapsed after allogeneic stem cell transplant for Hodgkin's Lymphoma or non-Hodgkin's Lymphoma (Group B)
* Life expectancy of greater than or equal to 6 weeks
* No severe intercurrent infection
* Patient, parent/guardian able to give informed consent
* Donor must be HIV negative (if autologous product used - patient must be HIV negative)
* Bilirubin less than or equal to 3x normal
* AST less than or equal to 5x normal
* Hgb higher than 8.0 g/L
* Creatinine less than or equal to 2x normal for age
* Patients should have been off other investigational therapy including T cells therapies for one month prior to entry in this study
* Karnofsky score of over or equal to 50
* No evidence of GVHD >Grade II at time of enrollment
* Female patients with reproductive capacity must have a negative pregnancy test

Exclusion Criteria:

* Patient, parent/guardian unable or unwilling to give informed consent
* Pregnant women
* Patients with a Karnofsky score of < 50
* Patients with a severe intercurrent infection
* Patients with a life expectancy of <6 weeks
* Patients with a bilirubin of more than 3x normal. AST of more than 5x normal
* Patients with a creatinine of more than 2x normal for age
* GVHD greater than Grade II at time of enrollment
* Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom

Note: Patients who would be excluded from the protocol strictly for laboratory abnormalities can be included at the investigator's discretion after approval by the CCGT Protocol Review Committee and the FDA reviewer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-10; Primary Completion 2006-02 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Adverse event data per patient | 6 weeks
  To determine the safety of autologous/syngeneic or allogeneic LMP-2 specific cytotoxic T-lymphocytes (CTL) in combination with CD45 monoclonal antibody (Mab) in patients with EBV positive Hodgkin's disease (HD) or non-Hodgkin's lymphoma (NHL).

SECONDARY OUTCOMES:
Survival of CTLs | up to 8 weeks
  Obtain information on expansion, persistence and anti-tumor effects of (CTL) given after lymphodepletion with CD45 monoclonal antibody (Mab) in patients with EBV positive Hodgkin's disease or non-Hodgkin's lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas